CLINICAL TRIAL: NCT04866017
Title: A Phase 3, Randomized, Open-Label Study to Compare Ociperlimab (BGB-A1217) Plus Tislelizumab (BGB-A317) Versus Durvalumab in Patients With Locally Advanced, Unresectable, PD-L1-Selected Non-Small Cell Lung Cancer Whose Disease Has Not Progressed After Concurrent Chemoradiotherapy
Brief Title: A Study to Compare Ociperlimab Plus Tislelizumab Versus Durvalumab Following Concurrent Chemoradiotherapy (cCRT) in Participants With Stage III Unresectable Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This decision was conducted by the sponsor and not driven by safety concerns as no new safety signals have been observed in the ociperlimab program.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-A1217-301; 2020-004656-14 (EudraCT Number); AdvanTIG-301 (Other: BeiGene)
Record Dates: First submitted 2020-10-28; First posted 2021-04-29 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; durvalumab; Drug Therapy; Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ociperlimab + Tislelizumab + cCRT (Experimental): Participants enrolled under PA1 recieved two cycles of ociperlimab combined with tislelizumab and cCRT, followed by ociperlimab combined with tislelizumab up to 1 year after the cCRT phase
  Interventions: Drug: Tislelizumab; Drug: Ociperlimab; Drug: Chemotherapy; Radiation: Radiotherapy
- Tislelizumab + cCRT (Experimental): Participants enrolled under PA1 recieved two cycles of tislelizumab combined with cCRT, followed by tislelizumab up to 1 year after the cCRT phase
  Interventions: Drug: Tislelizumab; Drug: Chemotherapy; Radiation: Radiotherapy
- cCRT followed by Durvalumab (Experimental): Participants enrolled under PA1 recieved two cycles of cCRT, followed by durvalumab to 1 year after the cCRT phase
  Interventions: Drug: Durvalumab; Drug: Chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — 200 mg intravenously every three weeks
  Other Names: BGB-A317
  Arms: Ociperlimab + Tislelizumab + cCRT; Tislelizumab + cCRT
Drug: Durvalumab — 10 milligrams per kilogram (mg/kg) intravenously once every 2 weeks (or 1500 mg intravenously once every 4 weeks where the dosage has been approved by a local health authority)
  Arms: cCRT followed by Durvalumab
Drug: Ociperlimab — 900 milligrams (mg) intravenously every three weeks
  Other Names: BGB-A1217
  Arms: Ociperlimab + Tislelizumab + cCRT
Drug: Chemotherapy — The chemotherapy regimen for the study treatment was selected at the investigator's discretion and may include one of the following options:
  * Cisplatin (50 mg/m²) on days 1 to 5 of each cycle, combined with etoposide (50 mg/m²) on days 1 and 8, both administered intravenously for 2 cycles. Each cycle was 28 days.
  * Carboplatin (AUC 2) weekly for 6 weeks, combined with paclitaxel (40-50 mg/m²) weekly for 6 weeks, both administered intravenously.
  * Cisplatin (75 mg/m²) combined with pemetrexed (500 mg/m²) on day 1 of each cycle, administered intravenously for 2 cycles. Each cycle was 21 days.
  * Carboplatin (AUC 5) combined with pemetrexed (500 mg/m²) on day 1 of each cycle, administered intravenously for 2 cycles. Each cycle was 21 days.
  The pemetrexed plus platinum regimen was only for participants with non-squamous histology.
  Other Names: Concurrent Chemoradiotherapy (cCRT)
Radiation: Radiotherapy — All participants recieved radiotherapy using either a standardized 3-dimensional conformal radiotherapy technique, or intensity modulated radiotherapy (IMRT) on a linear accelerator delivering a beam energy of ≥ 6 MV. The total dose of radiotherapy was 60 Gy, administered in 30 once-daily fractions of 2 Gy and 5 fractions per week for 6 weeks.
  Other Names: Concurrent Chemoradiotherapy (cCRT)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ociperlimab in combination with tislelizumab compared to durvalumab in adults with stage III unresectable PD-L1-selected non-small cell lung cancer whose disease has not progressed after cCRT.

DETAILED DESCRIPTION:
The study initiated with Protocol Amendment 1.0 (PA 1; dated on 16 April 2021). In April 2022 Protocol Amendment 2 (PA 2) was implemented. In PA 1, participants with newly diagnosed, histologically confirmed, unresectable locally advanced NSCLC and evaluable PD-L1 expression all comers were enrolled; cCRT was given within the study. In PA 2, the enrollment of the target population was revised into participants with unresectable locally advanced NSCLC whose disease has not progressed after definitive, platinum-based cCRT and with PD-L1 expression on ≥ 1% of tumor cells as assessed by the central lab; cCRT was given outside of the study.

After implementation of PA 2, participants who were randomized under PA 1 were given the option to continue assigned study treatment or to discontinue assigned treatment and begin standard of care treatment outside of the study. Participants enrolled under PA 1 were excluded from the primary and secondary analysis specified by PA 2.

This study was subsequently terminated by the Sponsor prior to enrollment of any participants under PA 2.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
2. Participant has histologically or cytologically confirmed, locally advanced, unresectable Stage III NSCLC (AJCC Cancer Staging Manual 2017, derived from IASLC) prior to initiation of cCRT.
3. Participant must have completed at least 2 cycles of platinum-based chemotherapy concurrent with radiotherapy
4. Participants must have not experienced PD following definitive, platinum-based cCRT.
5. Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Participants must have adequate organ function
7. Agree to provide archival tissue (formalin-fixed paraffin-embedded block containing tumor [preferred] or approximately 6 to 15 freshly cut unstained slides) or fresh biopsy obtained prior to cCRT (if archival tissue is not available) for prospective central evaluation of PD-L1 levels and retrospective analysis of other biomarkers.

Key Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, TIGIT, or any other antibody or drugs specifically targeting T-cell co-stimulation or checkpoint pathways.
2. Diagnosed with NSCLC that harbors an epidermal growth factor receptor (EGFR) sensitizing mutation, anaplastic lymphoma kinase (ALK) gene translocation, ROS1 gene translocation or RET gene rearrangement.
3. Participants who received systemic anticancer treatment besides the specified cCRT.
4. Any unresolved toxicity CTCAE > Grade 2 from the prior cCRT.
5. Active autoimmune diseases or history of autoimmune diseases that may relapse.
6. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone [in Japan, prednisolone] or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study treatment.
7. Infection (including tuberculosis infection, etc) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days before the first dose of study treatment.

Note: Antiviral therapy is permitted for participants with chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

NOTE: Other protocol Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- XCancer/Centeral Care Center, Bolivar, Missouri, United States
- Australia (7):
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Cabrini Hospital, Malvern, Victoria
  - Gold Coast University Hospital, Gold Coast
  - Hollywood Private Hospital, Perth
- China (20):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hunan Cancer Hospital - GCP Office, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital and Institute, Shandong First Medical University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - Changzhou Cancer Hospital, Changzhou
  - Jieyang People'S Hospital (Jieyang Affiliated Hospital, Sun Yat-Sen University ), Jieyang
- Spain (3):
  - Hospital Universitario Fundación Jiménez Díaz, Alcorcón, Madrid
  - Instituto Oncologico Dr. Rosell, Barcelona
  - Ico Girona, Girona
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in Taiwan, China, Spain , United States, and Australia. The first participant was consented on June 17th, 2021, and the last participant completed on October 17th, 2023. The decision to terminate the study was made on July 11th, 2023.
Pre-assignment Details: This study was initiated under Protocol Amendment (PA) 1. PA 2 was subsequently implemented; however, no participants were enrolled under PA 2 before the study was terminated. PA 2 changed the eligibility criteria, study treatment, study objectives and endpoints and excluded participants enrolled under PA 1 from analysis of the primary and secondary efficacy endpoint analyses.
Groups:
- Ociperlimab + Tislelizumab + cCRT: Participants enrolled in PA 1 received two cycles of ociperlimab (900 mg) and tislelizumab (200 mg) intravenously every three weeks, combined with concurrent chemoradiotherapy (cCRT). Chemotherapy regimens varied based on investigator discretion, including options such as cisplatin with etoposide, carboplatin with paclitaxel, or platinum-based regimens with pemetrexed for non-squamous histology; alongside radiotherapy. After the cCRT phase, participants continued ociperlimab and tislelizumab treatment for up to one year.
- Tislelizumab + cCRT: Participants in PA 1 received two cycles of tislelizumab (200 mg) intravenously every three weeks, combined with concurrent chemoradiotherapy (cCRT). The chemotherapy regimen was determined by the investigator and included options like cisplatin with etoposide, carboplatin with paclitaxel, or platinum-based regimens with pemetrexed for non-squamous histology; alongside radiotherapy. Following the cCRT phase, participants continued tislelizumab treatment for up to one year.
- cCRT Followed by Durvalumab: Participants in PA 1 received two cycles of concurrent chemoradiotherapy (cCRT), followed by durvalumab (10 mg/kg intravenously every 2 weeks, or 1500 mg every 4 weeks if locally approved). The chemotherapy regimen was chosen by the investigator and included options such as cisplatin with etoposide, carboplatin with paclitaxel, or pemetrexed with a platinum agent for non-squamous histology; alongside radiotherapy. After cCRT, participants continued durvalumab treatment for up to one year.
Period: Overall Study
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Started | 22 | 19 | 22
Treated | 22 | 18 | 22
Completed | 0 | 0 | 0
Not Completed | 22 | 19 | 22
Not completed — Study Terminated by Sponsor | 13 | 14 | 13
Not completed — Death | 8 | 4 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set is defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab | Total
Number analyzed (Participants) | 22 | 19 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.51) | 62.4 (9.27) | 64.1 (7.36) | 63.3 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 0 | 8
  Male | 19 | 14 | 22 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 18 | 15 | 18 | 51
  White | 4 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  China | 17 | 12 | 16 | 45
  Taiwan | 1 | 3 | 2 | 6
  Spain | 1 | 1 | 3 | 5
  United States | 2 | 1 | 1 | 4
  Australia | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: PFS is defined as the time from the date of randomization to the date of first documentation of disease progression as assessed by the IRC per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 or death, whichever occurred first.
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: The primary endpoint was specified in PA 2 and excludes participants enrolled under PA 1. No participants were enrolled under PA 2.
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomization until the date of death due to any cause
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: This secondary endpoint was specified in PA 2 and excludes participants enrolled under PA 1. No participants were enrolled under PA 2.
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) assessed by both the IRC and investigators per RECIST v1.1.
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: defined as the time from the first determination of a confirmed objective response assessed by both the IRC and investigators per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time to Death or Distant Metastasis (TTDM) as Assessed by the Investigator
Description: defined as the time from the date of randomization until the first date of distant metastasis assessed by both the IRC and investigators, or death. Distant metastasis is defined as any new lesion that is outside of the radiation field per RECIST v1.1 or proven by biopsy.
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Progression-Free Survival 2 (PFS2)
Description: defined as the time from randomization to the disease progression after next line of treatment, or death from any cause, whichever occurs first
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) determined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)
Time Frame: From first dose to 30 days after the last dose or initiation of a new anticancer therapy, whichever occured first; through study completion data cut-off date of October 17th, 2023 (maximum time on treatment was 16 months)
Population: The Safety Analysis Set included all randomized patients who received any dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 22 | 18 | 22
Participants
  TEAEs | 22 | 18 | 22
  SAEs | 11 | 8 | 8

8. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status
Description: Change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of participants with cancer. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline and Cycle 6 (Each cycle is 21 days)
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Assessed by Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13)
Description: Change from baseline in QLQ-CL13 scores for coughing, dyspnea, and chest pain. The QLQ-LC13 is a questionnaire that measures lung cancer-specific disease and treatment symptoms. It includes questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. A lower score indicates an improvement in symptoms.
Time Frame: Baseline and Cycle 6 (Each cycle is 21 days)
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Assessed by European Quality of Life-5 Dimensions (EQ-5D-5L)
Description: The EuroQol 5D-5L a descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the participant's health state.
Time Frame: Baseline and Cycle 6 (Each cycle is 21 days)
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Serum Concentration of Ociperlimab
Description: Serum concentrations of ociperlimab were measured for participants in the Ociperlimab + Tislelizumab + cCRT treatment group at predose (within 60 minutes before starting infusion) and postdose (within 30 minutes after the end of infusion). End of Treatment (EOT) visits occurred within 7 days after the date the investigator determined that study treatment would no longer be used, or before the initiation of a new anticancer treatment, whichever occurred first.
Time Frame: Predose at Day 1 of Cycles 1, 2, 5, 9, and 17; postdose on Day 1 of Cycles 1, 5 and EOT visit (Each Cycle was 21 days)
Population: The Pharmacokinetics (PK) Analysis Set includes all patients who receive any dose of any component of study drugs and for whom any postdose PK data are available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Groups:
- Ociperlimab + Tislelizumab + cCRT: Predose: Ociperlimab: 900 milligrams (mg) intravenously every three weeks. Predose was collected within 60 minutes before starting on Day 1 of Cycles 1, 2, 5, 9, and 17.
- Ociperlimab + Tislelizumab + cCRT: Postdose: Ociperlimab: 900 milligrams (mg) intravenously every three weeks. Postdose was collected within 30 minutes after end on infusion on Day 1 of Cycles 1 and 5, and at the EOT visit.
Arm/Group | Ociperlimab + Tislelizumab + cCRT: Predose | Ociperlimab + Tislelizumab + cCRT: Postdose
Number analyzed (Participants) | 22 | 22
ug/ml
  Cycle 1 Day 1 | 18 (NA) — Only one participant had a concentration level greater than the Lower Limit of Quantification (LLOQ). As a result, the variance and corresponding geometric coefficient of variation (CV) cannot be calculated. | 312 (45.82)
  Cycle 2 Day 1: number analyzed (Participants) | 20 | 0
  Cycle 2 Day 1 | 34.54 (63.19) |
  Cycle 5 Day 1: number analyzed (Participants) | 18 | 18
  Cycle 5 Day 1 | 74.86 (61.76) | 339.31 (38.21)
  Cycle 9 Day 1: number analyzed (Participants) | 12 | 0
  Cycle 9 Day 1 | 52.4 (82.40) |
  Cycle 17 Day 1: number analyzed (Participants) | 9 | 0
  Cycle 17 Day 1 | 81.35 (53.83) |
  End of Treatment: number analyzed (Participants) | 0 | 11
  End of Treatment |  | 94.94 (232.05)

12. Secondary Outcome: Serum Concentration of Tislelizumab for Participants in the Ociperlimab + Tislelizumab + cCRT Treatment Group
Description: Serum concentrations of tislelizumab were collected for participants in the Ociperlimab + Tislelizumab + cCRT treatment group at predose (within 60 minutes before starting infusion) and postdose (within 30 minutes after the end of infusion). End of Treatment (EOT) visits occurred within 7 days after the date investigator determined that study treatment would no longer be used, or before the initiation of a new anticancer treatment, whichever occurred first.
Time Frame: Predose at Day 1 of Cycles 1, 2, 5, 9, 17; postdose on Day 1 of Cycles 1 and 5, and EOT visit (each cycle was 21 days)
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Ociperlimab + Tislelizumab + cCRT: Predose: Tislelizumab 200 milligrams (mg) intravenously every three weeks. Predose was collected within 60 minutes before starting on Day 1 of Cycles 1, 2, 5, 9, and 17.
- Ociperlimab + Tislelizumab + cCRT: Postdose: Tislelizumab 200 milligrams (mg) intravenously every three weeks. Postdose was collected within 30 minutes after end on infusion on Day 1 of Cycles 1 and 5, and EOT visit.
Arm/Group | Ociperlimab + Tislelizumab + cCRT: Predose | Ociperlimab + Tislelizumab + cCRT: Postdose
Number analyzed (Participants) | 22 | 22
ug/mL
  Cycle 1 Day 1 | NA (NA) — No participants had concentration levels exceeding the LLOQ. | 72.20 (26.27)
  Cycle 2 Day 1: number analyzed (Participants) | 20 | 0
  Cycle 2 Day 1 | 15.91 (78.83) |
  Cycle 5 Day 1: number analyzed (Participants) | 18 | 18
  Cycle 5 Day 1 | 34.10 (49.67) | 97.08 (23.09)
  Cycle 9 Day 1: number analyzed (Participants) | 12 | 0
  Cycle 9 Day 1 | 30.22 (55.34) |
  Cycle 17 Day 1: number analyzed (Participants) | 9 | 0
  Cycle 17 Day 1 | 32.24 (156.53) |
  End of Treatment: number analyzed (Participants) | 0 | 11
  End of Treatment |  | 49.55 (89.19)

13. Secondary Outcome: Serum Concentration of Tislelizumab for Participants in the Tislelizumab + cCRT Treatment Group
Description: Serum concentrations of tislelizumab were collected for participants in the Tislelizumab + cCRT treatment group at predose (within 60 minutes prior to infusion initiation) and postdose (within 30 minutes after the completion of infusion). End of Treatment (EOT) visits occurred within 7 days after the date investigator determined that study treatment would no longer be used, or before the initiation of a new anticancer treatment, whichever occurred first.
Time Frame: Predose at Day 1 of Cycles 1, 2, 5, 9, and 17; postdose on Day 1 of Cycles 1 and 5, and EOT visit (Each Cycle is 21 days)
Population: PK Analysis Set; Tislelizumab concentration data are reported here for participants in the Tislelizumab + cCRT treatment group. Only participants with available data are included at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Tislelizumab: Predose: Tislelizumab 200 milligrams (mg) intravenously every three weeks. Predose was collected within 60 minutes before starting on Day 1 of Cycles 1, 2, 5, 9, 17, and EOT visit.
- Tislelizumab: Postdose: Tislelizumab 200 milligrams (mg) intravenously every three weeks. Postdose was collected within 30 minutes after end on infusion on Day 1 of Cycles 1 and 5
Arm/Group | Tislelizumab: Predose | Tislelizumab: Postdose
Number analyzed (Participants) | 17 | 17
ug/mL
  Cycle 1 Day 1 | NA (NA) — No participants had concentration levels exceeding the LLOQ. | 73.41 (18.53)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 0
  Cycle 2 Day 1 | 19.69 (27.01) |
  Cycle 5 Day 1: number analyzed (Participants) | 12 | 11
  Cycle 5 Day 1 | 37.64 (47.00) | 100.26 (29.25)
  Cycle 9 Day 1: number analyzed (Participants) | 12 | 0
  Cycle 9 Day 1 | 36.98 (39.63) |
  Cycle 17 Day 1: number analyzed (Participants) | 9 | 0
  Cycle 17 Day 1 | 41.29 (55.41) |
  End of Treatment: number analyzed (Participants) | 0 | 9
  End of Treatment |  | 40.18 (139.51)

14. Secondary Outcome: Immunogenic Responses to Ociperlimab as Assessed by the Detection of Treatment Emergent Anti-Drug Antibodies (ADAs)
Description: Defined as the sum of treatment-boosted and treatment-induced ADA participants as a proportion percentage of the ADA-evaluable participants population and is synonymous with 'ADA Incidence'. ADA samples were collected for participants randomized to Arm A (ociperlimab and tislelizumab)
Time Frame: Predose (within 60 minutes before dose) on Day 1 of Cycles 1, 2, 5, 9, 17, and the EOT Visit (Each cycle is 21 days). Maximum number of treatment cycles was 19
Population: The Immunogenicity Analysis Set includes all participants who received any dose of any component of study drugs and for whom both baseline antidrug antibody (ADA) and at least 1 postbaseline ADA result were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Ociperlimab + Tislelizumab + cCRT
Number analyzed (Participants) | 20
Participants | 0

15. Secondary Outcome: Immunogenic Responses to Tislelizumab as Assessed by the Detection of Treatment Emergent Anti-Drug Antibodies (ADAs)
Description: Defined as the sum of treatment-boosted and treatment-induced ADA participants as a proportion percentage of the ADA-evaluable participants population and is synonymous with 'ADA Incidence'. ADA samples were collected for participants randomized to Arm A (Ociperlimab + Tislelizumab + cCRT) and Arm B (Tislelizumab + cCRT)
Time Frame: Predose (within 60 minutes before dose) on Day 1 of Cycles 1, 2, 5, 9, 17, and the EOT Visit (Each cycle is 21 days, maximum number of treatment cycles was 19)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT
Number analyzed (Participants) | 20 | 17
Participants | 10 | 5

16. Secondary Outcome: Programmed Death-Ligand 1 (PD-L1) and T-cell Immunoreceptor With Ig and ITIM Domains (TIGIT) Expression in Archival and/or Fresh Tumor Tissues
Time Frame: From randomization through to the end of study, planned duration was 20 months
Population: as for outcome 2
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after the last dose or initiation of a new anticancer therapy, whichever occured first; through study completion data cut-off date of October 17th, 2023 (maximum time on treatment was 16 months)
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Ociperlimab + Tislelizumab + cCRT | Tislelizumab + cCRT | cCRT Followed by Durvalumab
All-Cause Mortality (participants affected / at risk) | 8/22 | 4/18 | 8/22
Serious Adverse Events (participants affected / at risk) | 11/22 | 8/18 | 8/22
Other Adverse Events (participants affected / at risk) | 22/22 | 18/18 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ociperlimab + Tislelizumab + cCRT (N=22) | Tislelizumab + cCRT (N=18) | cCRT Followed by Durvalumab (N=22)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ociperlimab + Tislelizumab + cCRT (N=22) | Tislelizumab + cCRT (N=18) | cCRT Followed by Durvalumab (N=22)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 10 (15) | 14 (20)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (4) | 2 (7) | 4 (9)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 1 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (3) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 4 (4)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (12) | 5 (9) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 7 (8) | 11 (18)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (5)
Asthenia (General disorders) | 4 (4) | 1 (1) | 5 (5)
Chest discomfort (General disorders) | 2 (3) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (3) | 1 (1) | 1 (2)
Chills (General disorders) | 1 (2) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 4 (5) | 2 (2)
Influenza like illness (General disorders) | 2 (4) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 3 (4)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 4 (7) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (4)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (5) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (3)
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 9 (10)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 5 (7)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (15) | 0 (0) | 6 (9)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (10) | 0 (0) | 4 (5)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3) | 2 (3) | 1 (1)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 1 (4) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (4) | 1 (2) | 2 (3)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (2) | 1 (3)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 1 (3) | 2 (4) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (4) | 3 (7) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (7) | 5 (5) | 6 (10)
Myoglobin blood increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 14 (31) | 5 (13) | 13 (29)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 8 (12) | 5 (6) | 10 (16)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 2 (2) | 4 (4)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 2 (2) | 4 (4)
Weight increased (Investigations) | 3 (6) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 15 (45) | 10 (25) | 13 (41)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 5 (7) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (14) | 1 (1) | 4 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (5) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (7) | 4 (6) | 3 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (6) | 6 (9) | 7 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1) | 3 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (6) | 5 (13) | 6 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 3 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 3 (3) | 1 (1)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (4) | 3 (4)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5) | 7 (7)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Since no participants were enrolled under PA 2, no analyses of the primary or secondary endpoints were conducted. Participants enrolled under PA 1 were excluded from the primary and secondary analyses outlined for PA 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04866017/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT04866017/SAP_001.pdf